CLINICAL TRIAL: NCT00703690
Title: A Multicenter, Double-Blind, Randomized, Placebo and Active-Controlled, Parallel Study to Evaluate the Lipid Altering Efficacy and Safety of MK0767 in Patients With Metabolic Syndrome and Dyslipidemia
Brief Title: MK0767 in Metabolic Syndrome-Dyslipidemia (0767-016)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-016; MK0767-016; 2007_641
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Metabolic X Syndrome Dyslipidemia
MeSH Terms: interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental): MK0767; 2.5 mg/day
  Interventions: Drug: MK0767
- 2 (Experimental): MK0767; 5mg/day
  Interventions: Drug: MK0767
- 3 (Experimental): MK0767; 10 mg/day
  Interventions: Drug: MK0767
- 4 (Active Comparator): fenofibrate 200 mg
  Interventions: Drug: Comparator: fenofibrate
- 5 (Placebo Comparator): Matching Placebo
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: MK0767 — MK0767 2.5, 5, and 10 mg/day supplied as tablets
  Arms: 1; 2; 3
Drug: Comparator: fenofibrate — fenofibrate 200 mg supplied as capsules
  Arms: 4
Drug: Comparator: Placebo (unspecified) — matching placebo will be supplied as tablets/capsules.
  Arms: 5

SUMMARY:
This is a clinical trial in patients with Metabolic Syndrome and Dyslipidemia to study the effects of MK0767 on triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Metabolic Syndrome and Dyslipidemia age 21 to 65
* Patients will be eligible for the study if their triglyceride levels are within protocol specified range and have at least 2 of the criteria for Metabolic Syndrome as defined by NCEP

Exclusion Criteria:

* Patients with a history of diabetes mellitus, partial ileal bypass, intolerant to fibric acid derivatives, requiring continuous oral corticosteroids, taking anti-seizure medications, documented coronary heart disease, renal insufficiency, proteinuria, viral hepatitis, cholelithiasis or other gallbladder disease, pancreatitis, neoplastic disease
* Patient is on cyclical estrogen medications
* Patient has taken lipid-lowering agents including fibric acid derivatives, bile acid sequestrants, HMG CoA reductase inhibitors and nicotinic acid derivatives within 8 weeks or probucol within 1 year of prior to visit 2

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2002-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
a dose-response will be seen across the doses of MK0767 and placebo in lowering fasting triglyceride. | After 12 weeks of treatment

SECONDARY OUTCOMES:
MK0767 will be safe and well tolerated | throughout study and at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC